CLINICAL TRIAL: NCT04533828
Title: Value of 68Ga-FAPI-04 PET/CT for Diagnosis and Prognostic Evaluation in Liver Fibrosis
Brief Title: 68Ga-FAPI PET/CT in Liver Fibrosis Patients
Acronym: GFAPILF
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPILF
Record Dates: First submitted 2020-08-22; First posted 2020-09-01 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Liver Fibrosis; Positron Emission Tomography
MeSH Terms: conditions — Liver Cirrhosis | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-04 PET/CT scanning (Experimental): Each subject receive a single intravenous injection of 68Ga-FAPI-04, and undergo PET/CT scanning within the specified time.
  Interventions: Drug: 68Ga-FAPI-04

INTERVENTIONS:
Drug: 68Ga-FAPI-04 — Each subject receive a single intravenous injection of 68Ga-FAPI-04, and undergo PET/CT scanning within the specified time.

SUMMARY:
To evaluate the potential value of 68Ga-FAPI-04 positron emission tomography/computed tomography (PET/CT) for the diagnosis and prognosis in liver fibrosis disease.

DETAILED DESCRIPTION:
Subjects with liver fibrosis underwent 68Ga-FAPI-04 PET/CT scanning. Liver fibrosis lesion uptake was quantified by the maximum standard uptake value (SUVmax). Subjects also received the conventional clinical assessment for liver fibrosis, such as transient elastography (TE) and blood biochemical indexes (BBI) testing. The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga-FAPI-04 PET/CT, TE and BBI were calculated and compared to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or order)
* patients with suspected or new diagnosed or previously treated liver fibrosis (supporting evidence may include TE, BBI, MRI, CT and pathology report)
* patients who had scheduled 68Ga-FAPI-04 PET/CT scan
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee

Exclusion Criteria:

* patients without liver fibrosis lesions
* patients with pregnancy
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 68Ga-FAPI-04 for each target lesion of subject or suspected liver fibrosis.

SECONDARY OUTCOMES:
Liver stiffness measurement (LSM) | 30 days
  Liver stiffness measurement (LSM) of transient elastography (TE) for each subject.
Blood biochemical indexes (BBI) testing | 30 days
  APRI (Aspartate aminotransferase to Platelet Ratio Index) and FIB-4 (Fibrosis-4) were calculated through blood biochemical indexes (BBI) testing for each subject.
  APRI = (AST)/(PLT)×100, FIB-4 = (Age×AST)/(PLT)×(ALT )^(1/2). ALT (Alanine transaminase), AST (Aspartate transaminase) and PLT (Platelets) counts were obtained from BBI testing.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No